CLINICAL TRIAL: NCT06776549
Title: Hypothermia Versus Normothermia After Extracorporeal Cardiopulmonary Resuscitation for Out-of-hospital Cardiac Arrest: A Cluster Randomized Trial (SAVE-J NEUROTHERM Trial)
Brief Title: Hypothermia Versus Normothermia After Extracorporeal Cardiopulmonary Resuscitation for Out-of-hospital Cardiac Arrest
Acronym: J-NEURO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kagawa University (Other)
Responsible Party: Principal Investigator, Akihiko Inoue, Principal Investigator, Kagawa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: j-neuro
Record Dates: First submitted 2025-01-03; First posted 2025-01-15 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-12

CONDITIONS: Out-of-hospital Cardiac Arrest (OHCA); ECMO Treatment; Temperature; Post Cardiac Arrest Syndrome
Keywords: Cardiac arrest; Out-of-hospital cardiac arrest (OHCA); Extracorporeal cardiopulmonary resuscitation (ECPR); Temperature control; Post cardiac arrest syndrome (PCAS)
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Post-Cardiac Arrest Syndrome; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normothermia (Active Comparator): Temperature control at 36 °C
  Interventions: Procedure: Temperature control
- Hypothermia (Experimental): Temperature control at 33-34 °C
  Interventions: Procedure: Temperature control

INTERVENTIONS:
Procedure: Temperature control — Procedure: Temperature control at 33-34 °C In the hypothermia group, patients receiving ECPR will be immediately cooled to 33ºC-34ºC with ECMO using a heat exchanger. After reaching this targeted temperature, the maintenance phase will start, and the target temperature will be kept at 33ºC-34°C. The maintenance phase will end 24 h after reaching this targeted temperature. Subsequently, rewarming to 36ºC-37ºC will be conducted in 24 h. After the rewarming, the temperature will be kept in the range of 36ºC-37.5ºC for 24 h after rewarming or until the end of ECMO, and should not exceed 37.5ºC. Other interventions, such as sedation, administration of neuromuscular blocking agents, antipyretics, and catecholamines, as well as mechanical circulatory support, are optional and performed at the patient's discretion.
  Arms: Hypothermia
Procedure: Temperature control — Procedure: Temperature control at 36 °C In the normothermia group receiving ECPR, the temperature of 36ºC will be immediately reached with ECMO using a heat exchanger. After reaching this targeted temperature, the maintenance phase will start, and the target temperature will be maintained at 36ºC. The maintenance phase will end 24 h after reaching this targeted temperature. Then, rewarming to 36ºC-37ºC will be conducted in 24 h. After the rewarming, the temperature will be kept in the range of 36ºC-37.5ºC for 24 h after rewarming or until the end of ECMO, and should not exceed 37.5ºC. Other interventions, such as sedation, administration of neuromuscular blocking agents, antipyretics, and catecholamines, as well as mechanical circulatory support, are optional and performed at the patient's discretion.
  Arms: Normothermia

SUMMARY:
The SAVE-J NEUROTHERM trial is a cluster randomized trial that evaluated and compared the mortality risk, neurological outcomes, and adverse events between patients who underwent hypothermia and those who underwent normothermia after extracorporeal cardiopulmonary resuscitation for out-of-hospital cardiac arrest.

DETAILED DESCRIPTION:
Temperature control is a key neurointensive care for post-cardiac arrest patients. Although therapeutic hypothermia has been shown to be effective in the past, recent large randomized controlled trials have failed to demonstrate its efficacy. The international guidelines recommend temperature control under 37.7°C. However, the optimal temperature control, i.e., hypothermia versus normothermia, remains controversial. Additionally, randomized controlled trials that examined temperature control after extracorporeal cardiopulmonary resuscitation (ECPR) are lacking.

ECPR is a resuscitation technique using extracorporeal membrane oxygenation (ECMO) for refractory cardiac arrest. In ECPR patients, ECMO using a heat exchanger can more rapidly achieve the targeted temperature as compared to other temperature control devices. Early cooling to achieve hypothermia after resuscitation is expected to be more effective for neuroprotection in the injured brain. Thus, the investigators hypothesized that hypothermia would be effective in ECPR patients.

Furthermore, ECMO can stabilize the respiratory and circulatory status. Therefore, hypothermia, which may have side effects such as electrolyte abnormalities and arrhythmias, may be safely performed by ECMO. However, ECMO requires the administration of anticoagulants; therefore, it has the risk of hemorrhagic complications. Among patients receiving ECPR, bleeding is a common complication due to its relatively difficult procedure, considering the fact that emergent cannulation is performed under resuscitation. Additionally, CPR-related complications can also result in bleeding. These complications may be enhanced by hypothermia. Therefore, hypothermia after ECPR could contribute to a favorable outcome, but it could also cause bleeding.

The SAVE-J NEUROTHERM trial is a cluster randomized trial that evaluated and compared the mortality risk, neurological outcomes, and adverse events between out-of-hospital cardiac arrest (OHCA) patients who underwent hypothermia and normothermia after ECPR.

ELIGIBILITY:
Inclusion Criteria:

* OHCA
* Age of 18-75 years, known or estimated
* An initial cardiac arrest rhythm of ventricular fibrillation/pulseless ventricular tachycardia or pulseless electrical activity

Exclusion Criteria:

* ECMO initiated after sustained return of spontaneous circulation (ROSC) and patients with sustained ROSC before ECMO initiation
* OHCA of presumed non-cardiac etiology
* Time from emergency call or witnessed arrest to hospital arrival of >60 min
* Time from hospital arrival to ECMO initiation of >60 min
* Pre-hospital ECPR
* Unavailability of the ECMO heat exchanger for temperature control
* Glasgow Coma Scale score before temperature control of >8
* Core body temperature upon hospital arrival of ≤32ºC
* Surgical intervention before temperature control (e.g., surgical intervention for the primary disease or complications related to resuscitation/ECMO procedures)
* Do Not Attempt Resuscitation) order confirmed prior to temperature control
* Limitations in intensive care before temperature control
* Known cerebral performance category (CPC) of 3-4 before cardiac arrest
* Known chronic obstructive pulmonary disease with home oxygen therapy
* Known or suspected pregnancy
* Concomitant illness, such as malignancy, shortens life expectancy (180-day survival unlikely)
* Consent not obtained or withdrawn by the participant or surrogate
* Other reasons, physician's decision not to enroll the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | At discharge (approximately 25 days)

SECONDARY OUTCOMES:
Survival | At 30 days, 90 days, and 1 year after admission
Neurological function: Cerebral performance categories (CPC) | At discharge (approximately 25 days), 30 days, 90 days, and 1 year after admission
  The range of cerebral performance category (CPC) score is from 1 (normal/good cerebral function) to 5 (brain death or death). The higher the score, the worse the outcome.
  A favorable neurological outcome was defined as a CPC of 1-2, whereas an unfavorable outcome was defined as a CPC of 3-5
Adverse events | During the intensive care unit stay, an average of 2 weeks
  Adverse events during intensive care unit stay (arrhythmia, bleeding, pneumonia, and bacteremia)

CONTACTS AND LOCATIONS:
Overall Officials: Akihiko Inoue, Principal Investigator — Hyogo Emergency Medical Center; Yasuhiro Kuroda, Study Chair — Kagawa University; Toru Hifumi, Study Chair — Kyorin University School of Medicine; Tetsuya Sakamoto, Study Director — Teikyo University; Naoaki Ichihara, Study Director — Osaka University
Locations (28):
- Japan (28):
  - Kurume University Hospital, Kurume, Fukuoka
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Prefectural Kakogawa Medical Center, Kakogawa, Hyōgo
  - Hyogo Emergency Medical Center, Kobe, Hyōgo
  - Toyooka Public Hospital, Toyooka, Hyōgo
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Oshima Prefectural Hospital, Amami, Kagoshima-ken
  - Ebina General Hospital, Ebina, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Kyoto Second Red Cross Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Sendai Medical Center, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Tsuyama Chuo Hospital, Tsuyama, Okayama-ken
  - Okinawa Prefectural Nanbu Medical Center & Children's Medical Center, Shimajiri-gun, Okinawa
  - Osaka Saiseikai Senri Hospital, Suita, Osaka
  - Saitama Red Cross Hospital, Saitama, Saitama
  - Tottori Prefectural Central Hospital, Tottori-shi, Tottori
  - St. Luke's International Hospital, Tokyo
  - Institute of Science Tokyo Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Japanese Red Cross Musashino Hospital, Tokyo
  - Tokyo Metropolitan Tama Medical Center, Tokyo
  - National Hospital Organization Disaster Medical Center, Tokyo